CLINICAL TRIAL: NCT03954938
Title: Influence of Craving Manipulation on Cocaine Self-Administration
Brief Title: Behavioral Effects of Drugs (Inpatient): 38
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19
Sponsor: William Stoops (Other)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED In 38
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Cocaine Use, Unspecified
MeSH Terms: interventions — Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Neutral-Look (Sham Comparator): Subjects will be instructed to look at cocaine associated images and respond naturally.
  Interventions: Behavioral: Craving Manipulation; Drug: Cocaine; Drug: Placebo
- Positive (Experimental): Subjects will be instructed to look at cocaine associated images and anticipate the positive aspects of engaging with the items shown.
  Interventions: Behavioral: Craving Manipulation; Drug: Cocaine; Drug: Placebo
- Negative (Active Comparator): Subjects will be instructed to look at cocaine associated images and anticipate the negative aspects of engaging with the items shown.
  Interventions: Behavioral: Craving Manipulation; Drug: Cocaine; Drug: Placebo

INTERVENTIONS:
Behavioral: Craving Manipulation — Craving will be manipulated based on instructions about cocaine associated images shown to subjects.
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined based on the craving manipulation condition.
Drug: Placebo — The pharmacodynamic effects of placebo will be determined based on the craving manipulation condition.

SUMMARY:
The specific aim of this project is to demonstrate that the decisional analysis/craving regulation aspects of CBT reduce cocaine self-administration in subjects with cocaine use disorder through diminished craving responses. Thirty non-treatment seeking human subjects meeting diagnostic criteria for cocaine use disorder will complete an outpatient, crossover, placebo-controlled study consisting of 1 practice and 9 experimental sessions. In each experimental session, the reinforcing effects of intranasal cocaine will be determined under one of three regulation of craving conditions that simulate CBT decisional analysis (i.e., negative instruction, positive instruction or a neutral "look" condition). After sampling the dose of cocaine available in each session, subjects will complete the craving manipulation assigned to that session, they will then rate their craving and finally they will have the opportunity to earn the sampled dose in a progressive-ratio procedure. We hypothesize that focusing on the negative effects of cocaine use will decrease craving and reduce cocaine self-administration relative to the positive and "look" conditions, and that craving will be positively correlated with self-administration outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance use disorder that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3x3 fully factorial crossover study with 9 conditions tested in random order in each completing subject. The factors are cocaine dose (0, 40, 80 mg) and craving manipulation (positive [anticipate positive aspects of consuming cocaine], negative [anticipate negative aspects of consuming cocaine], neutral [respond naturally]). Each of these conditions was combined (e.g., 0 mg cocaine with positive craving manipulation).
Groups:
- BED IN 38: Within subjects study assessing three craving manipulations and three cocaine doses.
Period: Overall Study
Arm/Group | BED IN 38
Started | 5
Positive-80 mg Cocaine | 5
Look-80 mg Cocaine | 5
Positive-40 mg Cocaine | 4
Look-0 mg Cocaine | 4
Positive-0 mg Cocaine | 3
Look-40 mg Cocaine | 3
Negative-0 mg Cocaine | 3
Negative-40 mg Cocaine | 3
Negative-80 mg Cocaine | 2
Completed | 2
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Completing subjects
Groups:
- Completing Subjects: Subjects who completed the full study (i.e., completed all craving induction and cocaine dose conditions)
Arm/Group | Completing Subjects
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Cocaine Was Selected
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure (Stoops et al., 2010) in which subjects can make 5 choices for each available cocaine dose. Reinforcing effects were measured for each cocaine dose during across the craving manipulation conditions.
Time Frame: One test for each of the craving manipulations for placebo and each cocaine dose level over approximately two weeks of participation.
Population: Completing Subjects; Only data from completing subjects included due to within subjects design of the project.
Measure: Mean (Standard Error); unit: Times Cocaine Selected
Groups:
- Neutral-Look-0 mg Cocaine: Subjects were instructed to look at cocaine associated images and respond naturally.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Placebo: The reinforcing effects of placebo were determined based on the craving manipulation condition.
- Positive-0 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the positive aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Placebo: The reinforcing effects of placebo were determined based on the craving manipulation condition.
- Negative-0 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the negative aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Placebo: The reinforcing effects of placebo were determined based on the craving manipulation condition.
  Placebo: The pharmacodynamic effects of placebo will be determined based on the craving manipulation condition.
- Neutral-Look-40 mg Cocaine: Subjects were instructed to look at cocaine associated images and respond naturally.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 40 mg cocaine were determined based on the craving manipulation condition.
- Positive-40 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the positive aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 40 mg cocaine were determined based on the craving manipulation condition
- Negative-40 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the negative aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 40 mg cocaine were determined based on the craving manipulation condition
- Neutral-Look-80 mg Cocaine: Subjects were instructed to look at cocaine associated images and respond naturally.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 80 mg cocaine were determined based on the craving manipulation condition.
- Positive-80 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the positive aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 80 mg cocaine were determined based on the craving manipulation condition
- Negative-80 mg Cocaine: Subjects were instructed to look at cocaine associated images and anticipate the negative aspects of engaging with the items shown.
  Craving Manipulation: Craving was manipulated based on instructions about cocaine associated images shown to subjects.
  Cocaine: The reinforcing effects of 80 mg cocaine were determined based on the craving manipulation condition
Arm/Group | Neutral-Look-0 mg Cocaine | Positive-0 mg Cocaine | Negative-0 mg Cocaine | Neutral-Look-40 mg Cocaine | Positive-40 mg Cocaine | Negative-40 mg Cocaine | Neutral-Look-80 mg Cocaine | Positive-80 mg Cocaine | Negative-80 mg Cocaine
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Times Cocaine Selected | 0 (0) | 0 (0) | 0 (0) | 1.5 (1.5) | 1 (1) | 1.5 (0.5) | 1 (1) | 2 (2) | 2 (0)

2. Secondary Outcome: Cocaine Craving
Description: Cocaine craving was assessed using a 10 point craving questionnaire that asks subjects to rate how much they are craving cocaine at that moment. The minimum craving score is 0 (i.e., no craving), the maximum craving score is 10 (i.e., highest craving).
Time Frame: Measured for each of the craving manipulations for placebo and each cocaine dose level over approximately two weeks of participation.
Population: Completing Subjects; Only data from completing subjects analyzed due to within subjects design of the project.
Measure: Mean (Standard Error); unit: units on a 10 point scale
Arm/Group | Neutral-Look-0 mg Cocaine | Positive-0 mg Cocaine | Negative-0 mg Cocaine | Neutral-Look-40 mg Cocaine | Positive-40 mg Cocaine | Negative-40 mg Cocaine | Neutral-Look-80 mg Cocaine | Positive-80 mg Cocaine | Negative-80 mg Cocaine
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
units on a 10 point scale | 1.5 (.5) | 1 (1) | .5 (.5) | 1.5 (.5) | 2.5 (.5) | 1.5 (.5) | 1 (0) | 3 (1) | 1.5 (.5)

ADVERSE EVENTS:
Time Frame: Two weeks of study participation
Description: This is a crossover, factorial study in which all subjects were randomly assigned to experience 9 conditions in random order.
Groups:
- Positive-0 mg Cocaine: Participants instructed to respond positively to cocaine images and receive 0 mg cocaine
- Positive-40 mg Cocaine: Participants instructed to respond positively to cocaine images and receive 40 mg cocaine
- Positive-80 mg Cocaine: Participants instructed to respond positively to cocaine images and receive 80 mg cocaine
- Look-0 mg Cocaine: Participants instructed to respond naturally to cocaine images and receive 0 mg cocaine
- Look-40 mg Cocaine: Participants instructed to respond naturally to cocaine images and receive 40 mg cocaine
- Look-80 mg Cocaine: Participants instructed to respond naturally to cocaine images and receive 80 mg cocaine
- Negative-0 mg Cocaine: Participants instructed to respond negatively to cocaine images and receive 0 mg cocaine
- Negative-40 mg Cocaine: Participants instructed to respond negatively to cocaine images and receive 40 mg cocaine
- Negative-80 mg Cocaine: Participants instructed to respond negatively to cocaine images and receive 80 mg cocaine
Arm/Group | Positive-0 mg Cocaine | Positive-40 mg Cocaine | Positive-80 mg Cocaine | Look-0 mg Cocaine | Look-40 mg Cocaine | Look-80 mg Cocaine | Negative-0 mg Cocaine | Negative-40 mg Cocaine | Negative-80 mg Cocaine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4 | 0/3 | 0/5 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4 | 0/3 | 0/5 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4 | 0/3 | 0/5 | 0/3 | 0/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive-0 mg Cocaine (N=3) | Positive-40 mg Cocaine (N=4) | Positive-80 mg Cocaine (N=5) | Look-0 mg Cocaine (N=4) | Look-40 mg Cocaine (N=3) | Look-80 mg Cocaine (N=5) | Negative-0 mg Cocaine (N=3) | Negative-40 mg Cocaine (N=3) | Negative-80 mg Cocaine (N=2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; only completing subjects' data analyzed due to within subjects design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03954938/Prot_SAP_000.pdf